CLINICAL TRIAL: NCT04913766
Title: REstoring Mental Health Through COmmUnity-based Psychological (RECOUP-NY)
Brief Title: REstoring Mental Health Through COmmUnity-based Psychological Services in New York City
Acronym: RECOUP-NY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: The New School (Other); Duke University (Other); Human Sciences Research Council (Other Government)
Responsible Party: Principal Investigator, Brandon A Kohrt, MD, PhD, Professor, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH127767 (NIH)
Record Dates: First submitted 2021-06-03; First posted 2021-06-04 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Depression; Anxiety; Psychological Distress; PTSD
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will not be given information on what intervention services the participants are receiving.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Services as usual (Active Comparator): Persons screening positive for depression will be referred from community-based organizations. The referrals will be made to mental health specialists who will provide care based on their standard of care.
  Interventions: Behavioral: Services as Usual
- Problem Management Plus (Experimental): Persons screening positive for depression will be offered Problem Management Plus delivered by community based organization staff.
  Interventions: Behavioral: Problem Management Plus

INTERVENTIONS:
Behavioral: Problem Management Plus — Five session psychological intervention focusing on problem management skills.
  Arms: Problem Management Plus
Behavioral: Services as Usual — Mental health services provided by a mental health specialists according to their standard practices of care
  Arms: Services as usual

SUMMARY:
The goal is to improve mental health. The study will evaluate the impact of community-based mental health services. Successful completion of this study will contribute to the National Institute of Mental Health Strategic Plan employing implementation science to maximize the public health impact of research for effectiveness and reach of mental health services in the United States.

DETAILED DESCRIPTION:
There is a need for delivery of psychological interventions by non-specialists when specialists are unable to meet the service demand. In the United States, training staff at community-based organizations to deliver psychological support has been highlighted as a way to increase availability of mental health services and increase access to mental health care, particularly for underserved populations. This study employs a mental health task-sharing model by partnering with community based organizations in New York City to train community based organizations staff without professional mental health training to deliver mental health services. This study examine the impact of community based organizations staff delivering mental health services to reduce mental health problems. This study is a cluster randomized control trial in New York City comparing Services as Usual arm and delivery of mental health services with Problem Management Plus (Intervention arm) among participating community based organizations. The target condition will be general psychological distress. This study will evaluate mental health outcomes populations served by community based organizations integrating Problem Management Plus into their other activities compared to community based organizations delivering services as usual. This study will evaluate implementation science outcomes to inform policy recommendations for of community-based delivery of psychological interventions. Successful completion of these aims will contribute to the 2020 National Institute of Mental Health Strategic Plan. Specifically, a) employing implementation science to maximize the public health impact of research for improving effectiveness and reach of mental health services, b) strengthening research-practice partnerships to expedite adoption, sustained implementation, and continuous improvement of evidence-based mental health services, and c) developing innovative service delivery models to dramatically improve outcomes of mental health services.

ELIGIBILITY:
Inclusion Criteria:

* Persons with Patient Health Questionnaire 4 scores equal to or above 3
* Functional impairment associated with psychological distress

Exclusion Criteria:

* Acute suicide risk
* Patient Health Questionnaire 4 score below 3
* No functional impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Psychological Outcome Profiles Questionnaire; Unabbreviated scale title "Psychological Outcome Profiles questionnaire" | 20 weeks after baseline assessment
  4-item self-report questionnaire that is a personalized measure of psychological distress.

SECONDARY OUTCOMES:
Patient Health Questionnaire 9; Unabbreviated scale title "Patient Health Questionnaire 9" | 20 weeks after baseline assessment
  9-item self-report scale to assess symptoms of depression, minimum value=0, maximum value=27, higher scores mean greater depression symptoms
Generalized Anxiety Disorder 7; Unabbreviated scale title "Generalized Anxiety Disorder 7" | 20 weeks after baseline assessment
  7-item self-report scale to assess symptoms of depression, minimum value=0, maximum value=21, greater scores mean more anxiety symptoms
Posttraumatic Stress Disorder Checklist 5; Unabbreviated scale title "Posttraumatic Stress Disorder Checklist 5" | 20 weeks after baseline assessment
  8-item self-report scale for symptoms of posttraumatic stress disorder, minimum value=0, maximum value=24, greater scores mean more posttraumatic stress symptoms
World Health Organization Disability Assessment Schedule; Unabbreviated scale title "World Health Organization Disability Assessment Schedule" | 20 weeks after baseline assessment
  12-item self report scale for disability, minimum score=0, maximum score=48, greater scores mean more disability

OTHER OUTCOMES:
Reducing Tension Checklist, Unabbreviated title "Reducing Tension Checklist" | 10 weeks after baseline assessment
  10 items self-report scale for psychosocial skill use, minimum score=0, maximum score=30, greater scores mean more skill use
Intolerance of Uncertainty Scale-Short Form; Unabbreviated title "Intolerance of Uncertainty Scale-Short Form" | 10 weeks after baseline assessment
  12-item self-report of responses to uncertainty, ambiguous situations, and the future

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Kohrt, MD, PhD, Principal Investigator — George Washington University
Locations (1):
- New School, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data will be shared through National Institute of Mental Health Data Archive
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication of the primary outcome findings
Access Criteria: Standard access requirements for National Institute of Mental Health Data Archive